CLINICAL TRIAL: NCT07150988
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of HSK44459 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Phase II Efficacy and Safety Study of HSK44459 in Subjects With Moderate to Severe Plaque Psoriasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK44459-206
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK44459 dose level 1 (Experimental): HSK44459 dosage 1 oral administration
  Interventions: Drug: HSK44459 dose level 1
- HSK44459 dose level 2 (Experimental): HSK44459 dose level 2 oral administration
  Interventions: Drug: HSK44459 dose level 2
- Placebo control (Placebo Comparator): placebo oral administration
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HSK44459 dose level 1 — HSK44459 dose level 1 oral administration
  Arms: HSK44459 dose level 1
Drug: HSK44459 dose level 2 — HSK44459 dose level 2 orally administration
  Arms: HSK44459 dose level 2
Drug: placebo — placebo oral adminisitration
  Arms: Placebo control

SUMMARY:
The purpose of this study is to assess the efficacy and safety of HSK44459 administered orally for moderate to severe plaque psoriasis in adults.

DETAILED DESCRIPTION:
Patients with moderate to severe plaque psoriasis will be randomized into 3 cohorts (dose level 1, dose level 2 and placebo). Approximately 150 subjects will be enrolled. This study includes an 16-week treatment Period, then a 4-week safety visit period.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand and voluntarily participate this trial, and sign the informed consent form;
* Age≥18 years, regardless of gender;
* Plaque psoriasis;
* A candidate for systemic therapy;
* Agree to use a highly effective method(s) of from the signing of the informed consent form to 3 months post-treatment.

Exclusion Criteria:

* Can not discontinue the prohibited medications specified in the protocol before the first dose and throughout the entire study period;
* Laboratory abnormalities with clinical significance;
* Forms of psoriasis other than chronic plaque-type;
* Presence of other dermatological or autoimmune diseases;
* Presence of active infection requiring systemic therapy;
* Has undergone or plans to undergo major surgery;
* History of cardiovascular or cerebrovascular diseases;
* History of suicide attempts or major psychiatric disorders;
* History of malignant tumors;
* History of gastrointestinal surgery or diseases that may have impact on the study;
* History of drug abuse, illicit drug use, or alcohol abuse;
* History of severe drug allergies;
* Pregnant or lactating women;
* Subjects with any other factor considered by the investigator to be ineligible for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-26 (Estimated); Primary Completion 2026-11-06 (Estimated); Study Completion 2026-11-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who have ≥75% reduction in PASI (PASI-75). | 16 weeks
  The proportion of subjects who have a reduction of 75% or more from baseline in the psoriasis area-and-severity index score (PASI 75) at week 16.

SECONDARY OUTCOMES:
Proportion of subjects achieving an IGA score of clear 0 or 1 with ≥2 point reduction from baseline. | 2, 4, 8, 12 and 16 weeks
  Proportion of subjects achieving an IGA score of clear 0 or 1 with ≥2 point reduction at week 2, 4, 8, 12 and 16 from baseline.
Proportion of subjects who have ≥75% reduction in PASI (PASI-75). | 2, 4, 8 and 12 weeks
  The proportion of subjects who have a reduction of 75% or more from baseline in the psoriasis area-and-severity index score (PASI 75) at week 2, 4, 8 and 12.
Proportion of subjects who have ≥50% reduction in PASI (PASI-50). | 2, 4, 8, 12 and 16 weeks
  The proportion of subjects who have a reduction of 50% or more from baseline in the psoriasis area-and-severity index score (PASI-50 at week 2, 4, 8, 12 and 16.
Proportion of subjects who have ≥90% reduction in PASI (PASI-90). | 2, 4, 8, 12 and 16 weeks
  The proportion of subjects who have a reduction of 90% or more from baseline in the psoriasis area-and-severity index score (PASI-90) at week 2, 4, 8, 12 and 16.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No